CLINICAL TRIAL: NCT03432858
Title: Endoscopic Carpal Tunnel Release, Infection Incidence, and Prophylactic Antibiotics: Indicated or Kick the Habit?
Brief Title: Preoperative Antibiotics for Carpal Tunnel Release Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Richard C Trevino, MD, Orthopedic Surgeon -WellSpan Orthopedics, WellSpan Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prophylactic Antibiotics: ESCR
Record Dates: First submitted 2018-02-06; First posted 2018-02-14 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Endoscopic Carpal Tunnel Release; Prophylactic Antibiotics
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Vancomycin; Cefazolin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Principal investigator, co-investigators, and participants are blinded to study intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin
- Cefazolin (Active Comparator)
  Interventions: Drug: Cefazolin
- Saline (Placebo Comparator)
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Vancomycin — Vancomycin - 1-gram dosing
  Arms: Vancomycin
Drug: Cefazolin — 2-gram dosing for patients <120 kg 3-gram dosing for patients 120 kg or greater
  Arms: Cefazolin
Drug: Saline Solution — Placebo
  Arms: Saline

SUMMARY:
This is a clinical trial to determine how effective antibiotics administered prior to endoscopic carpal tunnel release surgery are in preventing surgical site infections.

DETAILED DESCRIPTION:
Study participants will be randomized to a prophylactic IV antibiotic treatment arm (Vancomycin or Cefazolin) or a placebo IV saline solution. Subjects will be monitored following surgery for surgical site infections.

ELIGIBILITY:
Inclusion Criteria:

* High probability (>12 points) on the Carpal Tunnel-6 diagnostic aide
* Recommendation for carpal tunnel release
* Capable of providing informed consent/LAR to act on subject's behalf

Exclusion Criteria:

* Patients allergic to both penicillin/cephalosporins and vancomycin
* Patient immobilized with splint or cast
* Unwilling unable to provide informed consent
* Children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan Surgery and Rehab Hospital, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator 1: Vancomycin: 1-gram dosing
- Active Comparator 2: Cefazolin: 2-gram dosing for patients <120 kg 3-gram dosing for patients 120 kg or greater
- Placebo: Saline Solution: Placebo
Period: Overall Study
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Started | 12 | 83 | 89
Completed | 10 | 72 | 72
Not Completed | 2 | 11 | 17
Not completed — Protocol Violation | 2 | 1 | 9
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Procedure canceled/rescheduled | 0 | 9 | 6
Not completed — Required postop mobilization with splinting | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo | Total
Number analyzed (Participants) | 10 | 72 | 72 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 47 | 51 | 103
  >=65 years | 5 | 25 | 21 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (14.10) | 59.0 (15.37) | 55.8 (16.36) | 57.5 (15.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 46 | 47 | 100
  Male | 3 | 26 | 25 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 10 | 15
  Not Hispanic or Latino | 10 | 66 | 62 | 138
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 7
  White | 8 | 66 | 59 | 133
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 72 | 72 | 154

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infection
Description: Definitive diagnosis of infection of surgical site -wounds determined to be infected will be divided into superficial or deep infections and treated according to the standard of care at WellSpan health.
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Surgical Site Infection
Description: Definitive diagnosis of infection of surgical site -Definitive diagnosis of infection of surgical site -wounds determined to be infected will be divided into superficial or deep infections and treated according to the standard of care at WellSpan health.
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Diabetes Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infection that have diabetes
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Diabetes Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infection that have diabetes
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Surgical Site Infections That Use Tobacco
Description: Number of patients with surgical site infections that use tobacco products
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Surgical Site Infections That Use Tobacco
Description: Number of patients with surgical site infections that use tobacco products
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Chronic Obstructive Pulmonary Disease Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infections that have chronic obstructive pulmonary disease
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Chronic Obstructive Pulmonary Disease Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infections that have chronic obstructive pulmonary disease
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Anemia Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infections that have anemia
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Anemia Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infections that have anemia
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Peripheral Artery Disease Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infections that have peripheral artery disease
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Peripheral Artery Disease Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infections that have peripheral artery disease
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Surgical Site Infection and a History of Arthroplasty
Description: Number of patients with surgical site infections with history of arthroplasty
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Surgical Site Infection and History of Arthroplasty
Description: Number of patients with surgical site infections with history of arthroplasty
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Valvular Disease Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infections with valvular disease
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Valvular Disease Diagnosis and Surgical Site Infection
Description: Number of patients with surgical site infections with valvular disease
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Surgical Site Infection That Underwent Single Incision Endoscopic Carpal Tunnel Release
Description: Number of patients with surgical site infections with single incision ECTR
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Surgical Site Infection That Underwent Single Incision Endoscopic Carpal Tunnel Release
Description: Number of patients with surgical site infections with single incision ECTR
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Surgical Site Infection That Underwent Double Incision Endoscopic Carpal Tunnel Release
Description: Number of patients with surgical site infections with double incision ECTR
Time Frame: 2 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Surgical Site Infection That Underwent Double Incision Endoscopic Carpal Tunnel Release
Description: Number of patients with surgical site infections with double incision ECTR
Time Frame: 6 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 10 | 72 | 72
Participants | 0 | 0 | 0

21. Secondary Outcome: Time From Last Cortisone Injection
Description: For patients sustaining surgical site infection, the time from their last cortisone injection
Time Frame: 2 weeks post-operative
Population: No patients sustained surgical site infections and data were not collected for this Outcome Measure.
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Time From Last Cortisone Injection
Description: For patients sustaining surgical site infection, the time from their last cortisone injection
Time Frame: 6 weeks post-operative
Population: No patients sustained surgical site infections and data were not collected for this Outcome Measure.
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Acuity of Carpal Tunnel Syndrome
Description: For patients sustaining surgical site infection, the acuity of their carpal tunnel syndrome
Time Frame: 2 weeks post-operative
Population: No patients sustained surgical site infections and data were not collected for this Outcome Measure.
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Acuity of Carpal Tunnel Syndrome
Description: For patients sustaining surgical site infection, the acuity of their carpal tunnel syndrome
Time Frame: 6 weeks post-operative
Population: No patients sustained surgical site infections and data were not collected for this Outcome Measure
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks post procedure
Arm/Group | Active Comparator 1 | Active Comparator 2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/10 | 0/72 | 2/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator 1 (N=10) | Active Comparator 2 (N=72) | Placebo (N=72)
Pyogenic granuloma (Vascular disorders) | 0 | 0 | 1 (1)
Postoperative splinting (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) — Subject experienced wrist pain unrelated to wound or procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT03432858/Prot_SAP_000.pdf